CLINICAL TRIAL: NCT00606593
Title: Multicenter, Double-blind, Randomized, Placebo-controlled, 5-period, 5-treatment Crossover, Dose-finding Study to Evaluate the Efficacy and Safety of Oral Administration of ACT-078573 in Elderly Subjects With Chronic Primary Insomnia
Brief Title: Almorexant (ACT-078573) in Elderly Subjects With Chronic Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Midnight Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-057A201
Record Dates: First submitted 2008-01-04; First posted 2008-02-04 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Primary Insomnia
Keywords: insomnia; elderly; sleeplessness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — almorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- ABECD (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 oral capsules at 25 and 100 mg and matching placebo
- BCADE (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- CDBEA (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- DECAB (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- EADBC (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- DCEBA (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- EDACB (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- AEBDC (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- BACED (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo
- CBDAE (Experimental): 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Interventions: Drug: ACT-078573 and matching placebo

INTERVENTIONS:
Drug: ACT-078573 oral capsules at 25 and 100 mg and matching placebo — 5-period, 5-treatment crossover: sequences: ABECD, BCADE, CDBEA, DECAB, EADBC DCEBA, EDACB, AEBDC, BACED, CBDAE Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: ABECD
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: BCADE
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: CDBEA
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: DECAB
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: EADBC
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: DCEBA
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: EDACB
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: AEBDC
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: CBDAE
Drug: ACT-078573 and matching placebo — ACT-078573 oral capsules at 25 and 100 mg and matching placebo 5-period, 5-treatment crossover Where A = 200mg, B = 100 mg, C = 50 mg, D = 25mg, E = Placebo
  Arms: BACED

SUMMARY:
A 2-night polysomnography / 5-way cross-over study to evaluate the effect, safety and tolerability of oral administration of almorexant (ACT 078573) in elderly subjects with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Elderly subjects (> 64 years) with a diagnosis of primary insomnia.

Exclusion Criteria:

* History of any sleep disorder, or any Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) axis I disorder other than primary insomnia.
* Sleep apnea, or restless legs syndrome.
* Daytime napping of more than 1 hour per day.
* Important caffeine consumption, heavy tobacco use, alcohol or drug abuse within 2 years prior to the screening visit.
* Unwillingness to refrain from drugs, over-the-counter or herbal medication having an effect on sleep or behavior.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K. Walsh, PhD, Principal Investigator — Sleep Medicine and Research Center
Locations (21):
- United States (21):
  - Central Arkansas Research, Hot Springs, Arkansas
  - Pacific Sleep Medicine Services, Inc., Los Angeles, California
  - Pacific Sleep Medicine Services, Inc., San Diego, California
  - California Clinical Trials Medical Group, Inc., San Diego, California
  - PAB Clinical Research, Brandon, Florida
  - Miami Research Associates, Miami, Florida
  - OmniTrials, Naples, Florida
  - Broward Research Group & Sleep-Wake Disorders Center of South Florida, Pembroke Pines, Florida
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Clinical Neurophysiology Services, P.C., Troy, Michigan
  - Sleep Disorders & Research Center, Chesterfield, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Duke University, Durham, North Carolina
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio
  - Cleveland Clinic Health Systems, Cleveland, Ohio
  - Lynn Health Sciences Institute, Oklahoma City, Oklahoma
  - Sleep Disorders Center, Columbia, South Carolina
  - Sleep Medicine Associates P.A., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 242 subjects were screened at 18 centers in the United States and received single-blind placebo treatment. The first subject screening visit was 12 Dec 2007, the first subject was treated on 19 Dec 2007. 112 subjects were randomized, the first assigned double-blind treatment, was on 26 Dec 2007. Last subject, last clinic visit ended on 4 Apr 2008.
Pre-assignment Details: The study consisted of a 2-4-week screening phase on single-blind placebo, a 4-8-week treatment phase, and a 28 day safety follow-up. Subjects were randomized to one of 10 treatment sequences.
Groups:
- Treatment Sequence 200/100/P/50/25: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: almorexant (ACT-078573) 200 mg/ACT-078573 100 mg/Placebo/ACT-078573 50 mg/ACT-078573 25mg.
- Treatment Sequence 100/50/200/25/P: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 100 mg/ACT-078573 50 mg/ACT-078573 200 mg/ACT-078573 25 mg/placebo.
- Treatment Sequence 50/25/100/P/200: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 50 mg/ACT-078573 25 mg/ACT-078573 100 mg/placebo/ACT-078573 200 mg.
- Treatment Sequence 25/P/50/200/100: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 25 mg/placebo/ACT-078573 50 mg/ACT-078573 200 mg/ACT-078573 100 mg.
- Treatment Sequence P/200/25/100/50: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: placebo/ACT-078573 200 mg/ACT-078573 25 mg/ACT-078573 100 mg/ACT-078573 50 mg.
- Treatment Sequence 25/50/P/100/200: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 25 mg/ACT-078573 50 mg/placebo/ACT-078573 100 mg/ACT-078573 200 mg.
- Treatment Sequence P/25/200/50/100: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: placebo/ACT-078573 25 mg/ACT-078573 200 mg/ACT-078573 50 mg/ACT-078573 100 mg.
- Treatment Sequence 200/P/100/25/50: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 200 mg/placebo/ACT-078573 100 mg/ACT-078573 25 mg/ACT-078573 50 mg.
- Treatment Sequence 100/200/50/P/25: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 100 mg/ACT-078573 200 mg/ACT-078573 50 mg/placebo/ACT-078573 25 mg.
- Treatment Sequence 50/100/25/200/P: Study medication was administered in 5 treatment periods, each consisting of 2 consecutive treatment polysomnography (PSG) nights separated by 5-12 days of washout. Treatment consisted of two capsules containing study medication, orally administered on each of the 2 consecutive treatment nights. Treatments were administered in the following sequence: ACT-078573 50 mg/ACT-078573 100 mg/ACT-078573 25 mg/ACT-078573 200 mg/placebo.
Period: Overall Study
Arm/Group | Treatment Sequence 200/100/P/50/25 | Treatment Sequence 100/50/200/25/P | Treatment Sequence 50/25/100/P/200 | Treatment Sequence 25/P/50/200/100 | Treatment Sequence P/200/25/100/50 | Treatment Sequence 25/50/P/100/200 | Treatment Sequence P/25/200/50/100 | Treatment Sequence 200/P/100/25/50 | Treatment Sequence 100/200/50/P/25 | Treatment Sequence 50/100/25/200/P
Started | 11 (Randomized participants) | 11 (Randomized participants) | 11 (Randomized participants) | 11 (Randomized participants) | 12 (Randomized participants) | 11 (Randomized participants) | 11 (Randomized participants) | 11 (Randomized participants. One participant actually received the treatment sequence 200/P/100/ 50/25) | 12 (Randomized participants) | 11 (Randomized participants)
1st Double-blind Treatment | 11 | 11 | 11 | 11 | 12 | 11 | 11 | 11 | 12 | 11
2nd Double-blind Treatment | 11 | 11 | 11 | 10 | 12 | 11 | 10 | 9 | 12 | 11
3rd Double-blind Treatment | 11 | 11 | 10 | 10 | 11 | 11 | 10 | 9 | 12 | 11
4th Double-blind Treatment | 10 | 11 | 10 | 10 | 11 | 11 | 10 | 9 | 11 | 11
5th Double-blind Treatment | 10 | 11 | 9 | 10 | 11 | 11 | 10 | 9 | 11 | 11
Completed | 10 | 11 | 9 | 10 | 11 | 11 | 10 | 9 | 11 | 11
Not Completed | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0
Not completed — Withdrawal of consent | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative/Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patient Flow: The study consisted of a 2-4-week screening phase (including 2 consecutive screening polysomnography (PSG) nights on single blind placebo), a 4- to 8-week treatment phase, and a 28 day safety follow-up. The treatment phase immediately followed randomization and included 5 treatment periods, each consisting of 2 consecutive treatment PSG nights on the assigned study treatment separated by 5 to 12 days of washout. Subjects were randomized to one of 10 treatment sequences.
Arm/Group | Patient Flow
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Mean Wake Time After Sleep Onset (WASO)
Description: WASO was the time in minutes scored as wake between the onset of persistent sleep and lights on, where the onset of persistent sleep was the beginning of the first continuous 20 epochs (10 min) scored as non-wake.
  Mean values were calculated based on 2 treatment PSG nights. PSG nights identified as non-evaluable due to protocol violation were excluded. If a mean value could not be calculated because the value for 1 PSG night was missing or non-evaluable, the valid value for the other PSG night was used. If during a double-blind treatment period a valid PSG was performed but the WASO was missing (e.g., persistent sleep did not occur), the missing value was substituted with the highest value recorded for the subject during the study (single-blind period included).
Time Frame: 2 treatment nights
Population: Number of evaluable patients for this parameter in the per protocol set. Only subjects with all 5 valid values are included in this analysis.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Placebo: Two capsules containing placebo, orally administered on each of 2 consecutive nights
- ACT-078573 25 mg: Two capsules containing ACT-078573 25 mg, orally administered on each of 2 consecutive nights
- ACT-078573 50 mg: Two capsules containing ACT-078573 50 mg, orally administered on each of 2 consecutive nights
- ACT-078573 100 mg: Two capsules containing ACT-078573 100 mg, orally administered on each of 2 consecutive nights
- ACT-078573 200 mg: Two capsules containing ACT-078573 200 mg, orally administered on each of 2 consecutive nights
Arm/Group | Placebo | ACT-078573 25 mg | ACT-078573 50 mg | ACT-078573 100 mg | ACT-078573 200 mg
Number analyzed (Participants) | 100 | 100 | 100 | 100 | 100
minutes | 109.1 (36.0) | 98.7 (35.5) | 90.0 (35.7) | 77.7 (33.2) | 62.6 (27.5)
Statistical Analysis 1: Comparison: Placebo vs ACT-078573 25 mg; Test type: Superiority or Other; p = 0.0018, Linear model; Least square means treatment effect = -10.4, 95% CI 2-sided [-17.0 to -3.9]
Statistical Analysis 2: Comparison: Placebo vs ACT-078573 50 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = -19.2, 95% CI 2-sided [-25.7 to -12.6]
Statistical Analysis 3: Comparison: Placebo vs ACT-078573 100 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = -31.4, 95% CI 2-sided [-38.0 to -24.9]
Statistical Analysis 4: Comparison: Placebo vs ACT-078573 200 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = -46.5, 95% CI 2-sided [-53.3 to -39.9]

2. Secondary Outcome: Mean Total Sleep Time (TST)
Description: TST was the amount of actual sleep time measured in minutes scored as non-wake (i.e., sleep stage 1, 2, slow-wave sleep, or rapid eye movement (sleep)).
  Mean values were calculated based on 2 treatment PSG nights. PSG nights identified as non-evaluable by protocol violation were excluded. If a mean value could not be calculated because the value for 1 PSG night was missing or non-evaluable, the valid value for the other PSG night was used. If during a double-blind treatment period a valid PSG was performed but the TST was missing (e.g., the subject did not sleep or persistent sleep did not occur), the missing value was substituted with the worst value recorded for the subject during the study (single-blind period included).
Time Frame: 2 treatment nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | ACT-078573 25 mg | ACT-078573 50 mg | ACT-078573 100 mg | ACT-078573 200 mg
Number analyzed (Participants) | 100 | 100 | 100 | 100 | 100
minutes | 339.7 (43.2) | 353.8 (40.1) | 360.9 (41.7) | 374.2 (39.6) | 394.7 (34.6)
Statistical Analysis 1: Comparison: Placebo vs ACT-078573 25 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = 14.3, 95% CI 2-sided [7.4 to 21.2]
Statistical Analysis 2: Comparison: Placebo vs ACT-078573 50 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = 21.5, 95% CI 2-sided [14.6 to 28.4]
Statistical Analysis 3: Comparison: Placebo vs ACT-078573 100 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = 34.7, 95% CI 2-sided [27.8 to 41.6]
Statistical Analysis 4: Comparison: Placebo vs ACT-078573 200 mg; Test type: Superiority or Other; p < 0.0001, Linear model; Least square means treatment effect = 55.1, 95% CI 2-sided [48.2 to 62.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events and serious adverse events were collected during each treatment period. Each treatment period included up to 4 days after the last administration of study treatment.
Description: Safety population
Groups:
- Single-blind Placebo: Treatment administered during screening period
Arm/Group | Single-blind Placebo | Placebo | ACT-078573 25 mg | ACT-078573 50 mg | ACT-078573 100 mg | ACT-078573 200 mg
Serious Adverse Events (participants affected / at risk) | 0/112 | 1/107 | 0/106 | 0/106 | 0/106 | 0/108
Other Adverse Events (participants affected / at risk) | 5/112 | 12/107 | 12/106 | 10/106 | 11/106 | 10/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-blind Placebo (N=112) | Placebo (N=107) | ACT-078573 25 mg (N=106) | ACT-078573 50 mg (N=106) | ACT-078573 100 mg (N=106) | ACT-078573 200 mg (N=108)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Placebo (N=112) | Placebo (N=107) | ACT-078573 25 mg (N=106) | ACT-078573 50 mg (N=106) | ACT-078573 100 mg (N=106) | ACT-078573 200 mg (N=108)
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 4 | 1 | 2 | 2
HEADACHE (Nervous system disorders) | 2 | 2 | 0 | 3 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 1
FATIGUE (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
EYE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
EYE INFECTION VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
RHINITIS SEASONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
SEDATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
URETHRAL PAIN (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
EYE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other